CLINICAL TRIAL: NCT00319774
Title: Assessment of Hemocontrol Biofeedback System Efficiency on Long Term Blood Pressure Control, Nursing Interventions, and Quality of Life in Hemodialysis Patients: a Randomized Controlled Trial
Brief Title: Hemocontrol and Blood Pressure Control in Dialysis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Université de Montréal (Other)
Collaborators: Gambro Renal Products, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HC-01
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Last update posted 2006-04-27 (Estimated); Status verified 2003-09

CONDITIONS: End-Stage Renal Disease; Hemodialysis
Keywords: End-stage renal disease; Hemodialysis; Hypertension; Hypotension; Blood volume; Hypervolemia; Quality of life; Biofeedback system
MeSH Terms: conditions — Kidney Failure, Chronic; Hypertension; Hypotension; Edema

INTERVENTIONS:
Device: Hemocontrol Biofeedback System

SUMMARY:
Volume overload contributes significantly to the pathogenesis of hypertension in hemodialysis patients. The Hemocontrol(HC)system (Gambro), which automatically adjusts ultrafiltration rate and dialysate conductivity according to blood volume variations during dialysis, has been suggested to improve hemodynamic tolerance and thus facilitate fluid removal.

This randomized controlled trial was designed to compare the use of HC with standard hemodialysis to test the hypothesis that the use of the HC system may lower home blood pressure in comparison with standard hemodialysis as a primary endpoint. Secondary endpoints are a variation in the percentage of dialysis sessions requiring nurses' interventions for intra-dialytic hypotension and a change in the health-related quality of life of HD patients.

DETAILED DESCRIPTION:
Hypertension is a common problem in patients undergoing chronic maintenance hemodialysis (HD) with a reported prevalence of 50 to 90 % [Hörl, 2002]. As a major risk factor for cardiovascular disease, hypertension contributes to the high rate of morbidity and mortality in ESRD patients [Foley, 1996; Port, 1999]. For a majority of dialysis patients, volume overload (VO) plays a major role in the pathogenesis of hypertension [Fishbane, 1996; Rahman, 2000; Ventura, 1997] and removing excess volume can often normalize blood pressure [Fishbane, 1996]. Unfortunately, correcting VO frequently proves to be difficult because of hemodynamic instability during HD sessions. As much as 20 to 50% of dialysis patients present with symptoms of intradialytic hypotension (IDH) [Santoro, 2002]. IDH increases nursing work load and negatively affects the efficacy of dialysis and the quality of life of HD patients. Different measures are used to avoid IDH, such as limitation of salt and water intake, avoidance of antihypertensive medication before dialysis, utilization of low temperature dialysate, and modeling of ultrafiltration and/or dialysate conductivity. These measures often generate mixed results.

The Hemocontrol (HC) biofeedback system (Gambro®) has been reported to reduce hemodynamic instability and hypotensive episodes during hemodialysis [Basile, 2001; Begin, 2002; Ronco, 2000; Santoro, 1994; Santoro, 1998; Santoro, 2002; Wolkotte, 2002]. The HC system consists in a fully integrated biofeedback system that monitors and regulates blood volume contraction during hemodialysis through software-driven adjustments of ultrafiltration rate and dialysate conductivity. By improving hemodynamic tolerance during dialysis, the use of the HC system has been suggested to facilitate fluid removal and correction of VO, leading to improved control of hypertension.

The present randomized controlled trial was designed to test the hypothesis that the use of the HC system would lower home BP in comparison with standard hemodialysis as a primary endpoint. Secondary endpoints are a variation in the percentage of HD sessions requiring nurses' interventions and a change in the health-related quality of life of HD patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* chronic hemodialysis
* on renal replacement therapy > 3 months
* at least 3 dialysis sessions and 9 hours of therapy weekly
* willing to measure blood pressure at home
* able to sign an informed consent

Exclusion Criteria:

* anticipated change in renal replacement therapy
* anticipated transfer to another center
* planned renal transplantation
* enrollment in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2002-12; Study Completion 2003-07

PRIMARY OUTCOMES:
Difference from baseline to end of study in ambulatory blood pressure control

SECONDARY OUTCOMES:
Episodes of intra-dialytic hypotension requiring nursing interventions
Health-related quality of life (using the Kidney Disease and Quality of Life Short Form)

CONTACTS AND LOCATIONS:
Overall Officials: Francois Madore, MD, Principal Investigator — Faculty of Medicine, University of Montreal
Locations (1):
- Hopital du Sacre-Coeur de Montreal, Montreal, Quebec, Canada

REFERENCES:
- [Background] C. Déziel, M. Zellweger, R. Comeau, A. Valleau, S. Raymond-Carrier, F. Madore. Home Blood Pressure Management with Automated Blood Volume Regulation in Hemodialysis Patients: A Prospective Randomized Controlled Trial. J. Am. Soc. Nephrol. 15:594A, October 2004.
- [Background] C. Déziel, M. Zellweger, R. Comeau, M. Kerangueven, S. Raymond-Carrier, F. Madore. Hemodynamic Stability during Hemodialysis and Quality of Life with Automated Blood Volume Regulation: A Prospective Randomized Controlled Trial. J. Am. Soc. Nephrol. 15:47A, October 2004